CLINICAL TRIAL: NCT04932655
Title: A Four-way Crossover Food Effect and Bioequivalence Pharmacokinetic Study of Simufilam in Healthy Volunteers
Brief Title: Food Effect and Bioequivalence Study of Simufilam Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cassava Sciences, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PTI-125-05
Record Dates: First submitted 2021-05-19; First posted 2021-06-21 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Simufilam

STUDY DESIGN:
Intervention Model Description: Four-way crossover of Phase 3 tablets under fasted or high-fat or low-fat conditions and the Phase 2 tablet under fasted conditions. Subjects are randomized to a sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence A (Other): This arm received Phase 2 tablet fasted (Period 1), Phase 3 tablet fasted (Period 2), Phase 3 tablet after a high-fat meal (Period 3), and Phase 3 tablet after a low-fat meal (Period 4).
  Interventions: Drug: simufilam
- Sequence B (Other): This arm received Phase 3 tablet after a low-fat meal (Period 1), Phase 2 tablet fasted (Period 2), Phase 3 tablet fasted (Period 3), and Phase 3 tablet after a high-fat meal (Period 4).
  Interventions: Drug: simufilam
- Sequence C (Other): This arm received Phase 3 tablet fasted (Period 1), Phase 3 tablet after a high-fat meal (Period 2), Phase 3 tablet after a low-fat meal (Period 3), and Phase 2 tablet fasted (Period 4).
  Interventions: Drug: simufilam
- Sequence D (Other): This arm received Phase 3 tablet after a high-fat meal (Period 1), Phase 3 tablet after a low-fat meal (Period 2), Phase 2 tablet fasted (Period 3), and Phase 3 tablet fasted (Period 4).
  Interventions: Drug: simufilam

INTERVENTIONS:
Drug: simufilam — Simufilam 100 mg oral tablets: the Phase 3 oral tablet for the first 3 arms and the Phase 2 tablet for the 4th arm.
  Other Names: PTI-125

SUMMARY:
This study will compare the pharmacokinetics of the Phase 3 simufilam 100 mg oral tablet when taken fasted versus following a high-fat or low-fat meal. Additionally, the Phase 3 oral tablet will be compared to the Phase 2 oral tablet for bioequivalence under fasted conditions.

DETAILED DESCRIPTION:
This is a single-center, randomized, four-treatment, four-sequence crossover study in healthy volunteers to estimate the effect of food on the pharmacokinetics of simufilam following oral 100 mg Phase 3 oral tablets. Additionally, the relative bioavailability of the Phase 3 100 mg tablet will be compared to the earlier Phase 2 100 mg tablet in the fasted state. A total of twenty four (24) healthy volunteers (12 male and 12 female) will be enrolled into this study. Subjects will be randomly assigned to one of four treatment sequences (6 subjects/sequence).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, Ages ≥ 18 and ≤ 45 years
2. BMI of 18 - 30 Kg/m²
3. Informed consent form (ICF) signed by the subject
4. General health status acceptable for participation in the study as determined by medical history, review of current medication, physical examination, and laboratory results
5. Fluency (oral and written) in English
6. The patient must agree to comply with the drawing of blood samples for the PK assessments, laboratory assessments and plasma biomarkers
7. The subject is willing and able to remain at the study site for the duration of the study

Exclusion Criteria:

1. The subject has any relevant deviations from normal in physical examination, electrocardiogram (ECG), or clinical laboratory tests, as evaluated by the investigator.
2. The subject has had a clinically significant illness within 30 days of this study.
3. The subject has a history of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease.
4. Subject is taking prescription CNS medication.
5. The subject has used alcohol, grapefruit, grapefruit juice, caffeine or xanthinecontaining products 48 h before dosing or intends to use any of these products during the study.
6. The subject has a history of substance abuse or a current positive ethanol breath test or positive urine drug screen.
7. The subject has a positive serum hepatitis B surface antigen or positive HCV antibody test.
8. The subject has a positive HIV test.
9. The subject has a current positive urine cotinine test.
10. The subject has participated in another drug study in the past 30 days.
11. The subject has donated or lost a significant volume of blood (>450 mL) within 4 weeks of the study.
12. The subject is unwilling to reside in the study unit for the duration of the study or to cooperate fully with the investigator or site personnel.
13. Covid-19 infection within the past 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Bass, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials Phase I Unit, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (2.14) | 38.0 (3.52) | 30.3 (4.18) | 34.7 (7.09) | 33.7 (5.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 2 | 9
  Male | 4 | 5 | 2 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 4 | 1 | 10
  Not Hispanic or Latino | 2 | 5 | 2 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 1 | 4 | 11
  White | 4 | 2 | 4 | 1 | 11
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24
Height [Mean (Standard Deviation); unit: cm] | 172.08 (10.24) | 174.95 (6.37) | 168.70 (10.65) | 173.62 (14.43) | 172.34 (10.36)
Weight [Mean (Standard Deviation); unit: Kg] | 79.25 (11.70) | 75.77 (14.63) | 69.78 (15.92) | 80.58 (18.70) | 76.35 (15.02)
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 26.63 (1.85) | 24.62 (3.49) | 24.35 (3.51) | 26.45 (2.55) | 25.51 (2.93)

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: The maximum concentration determined directly from individual concentration-time data
Time Frame: 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fasted Phase 3 Simufilam: All subjects following Phase 3 simufilam 100 mg taken in a fasted state.
- Phase 3 High-fat Fed Simufilam: All subjects following Phase 3 simufilam 100 mg taken 30 min after the start of a high-fat meal.
- Phase 3 Low-fat Fed Simufilam: All subjects following Phase 3 simufilam 100 mg taken 30 min after the start of a low-fat meal.
- Fasted Phase 2 Simufilam: All subjects after taking the Phase 2 simufilam oral tablet in a fasted state.
Arm/Group | Fasted Phase 3 Simufilam | Phase 3 High-fat Fed Simufilam | Phase 3 Low-fat Fed Simufilam | Fasted Phase 2 Simufilam
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 698 (190) | 715 (156) | 755 (149) | 680 (193)
Statistical Analysis 1: Comparison: Fasted Phase 3 Simufilam vs Phase 3 High-fat Fed Simufilam; Test type: Equivalence — Two one-sided t test procedure used to compare test versus reference. Equivalence demonstrated if 90% CI within 80% to 125%; Test/Reference Ratio of Geometric Means = 103.22, 90% CI 2-sided [96.88 to 109.98]
Statistical Analysis 2: Comparison: Fasted Phase 3 Simufilam vs Phase 3 Low-fat Fed Simufilam; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Test/Reference Ratio of Geometric Means = 109.64, 90% CI 2-sided [102.9 to 116.82]
Statistical Analysis 3: Comparison: Fasted Phase 3 Simufilam vs Fasted Phase 2 Simufilam; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Test/Reference Ratio of Geometric Means = 102.90, 90% CI 2-sided [96.57 to 109.64]

2. Primary Outcome: AUClast
Description: Area under the curve to the time of the last quantifiable concentration, calculated using the linear trapezoidal method
Time Frame: 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Fasted Phase 3 Simufilam: All subjects following Phase 3 simufilam 100 mg tablet in a fasted state.
- Phase 3 High-fat Fed Simufilam: All subjects following Phase 3 simufilam 100 mg tablet taken 30 min after the start of a high-fat meal.
- Phase 3 Low-fat Fed Simufilam: All subjects following Phase 3 simufilam 100 mg tablet taken 30 min after the start of a low-fat meal.
- Fasted Phase 2 Simufilam: All subjects following Phase 2 simufilam 100 mg tablet taken in a fasted state.
Arm/Group | Fasted Phase 3 Simufilam | Phase 3 High-fat Fed Simufilam | Phase 3 Low-fat Fed Simufilam | Fasted Phase 2 Simufilam
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 3890 (1050) | 3810 (951) | 3830 (971) | 3860 (978)
Statistical Analysis 1: Comparison: Fasted Phase 3 Simufilam vs Phase 3 High-fat Fed Simufilam; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Test/Reference Ratio of Geometric Means = 98.47, 90% CI 2-sided [96.33 to 100.65]
Statistical Analysis 2: Comparison: Fasted Phase 3 Simufilam vs Phase 3 Low-fat Fed Simufilam; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Test/Reference Ratio of Geometric Means = 98.88, 90% CI 2-sided [96.74 to 101.07]
Statistical Analysis 3: Comparison: Fasted Phase 3 Simufilam vs Fasted Phase 2 Simufilam; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Test/Reference Ratio of Geometric Means = 100.32, 90% CI 2-sided [98.15 to 102.54]

3. Primary Outcome: AUCinf
Description: Area under the curve extrapolated to infinity; calculated as: AUCinf = AUClast + Clast/λz
Time Frame: 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Fasted Phase 3 Simufilam | Phase 3 High-fat Fed Simufilam | Phase 3 Low-fat Fed Simufilam | Fasted Phase 2 Simufilam
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 3980 (1130) | 3900 (1030) | 3930 (1050) | 3960 (1060)
Statistical Analysis 1: Comparison: Fasted Phase 3 Simufilam vs Phase 3 High-fat Fed Simufilam; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Test/Reference Ratio of Geometric Means = 98.50, 90% CI 2-sided [96.33 to 100.71]
Statistical Analysis 2: Comparison: Fasted Phase 3 Simufilam vs Phase 3 Low-fat Fed Simufilam; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Test/Reference Ratio of Geometric Means = 99.03, 90% CI 2-sided [96.85 to 101.26]
Statistical Analysis 3: Comparison: Fasted Phase 3 Simufilam vs Fasted Phase 2 Simufilam; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Test/Reference Ratio of Geometric Means = 100.25, 90% CI 2-sided [98.05 to 102.50]

ADVERSE EVENTS:
Time Frame: 8 days
Arm/Group | Fasted Phase 3 Simufilam | Phase 3 High-fat Fed Simufilam | Phase 3 Low-fat Fed Simufilam | Fasted Phase 2 Simufilam
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 4/24 | 3/24 | 2/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4.17% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasted Phase 3 Simufilam (N=24) | Phase 3 High-fat Fed Simufilam (N=24) | Phase 3 Low-fat Fed Simufilam (N=24) | Fasted Phase 2 Simufilam (N=24)
headache (Nervous system disorders) | 0 | 1 (1) | 1 (1) | 0
nausea (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
constipation (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0
abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0
dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0
auditory disorder (Ear and labyrinth disorders) | 1 (1) | 0 | 0 | 0
fatigue (General disorders) | 0 | 1 (1) | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0
diarrhoea (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 0
Lacrimal disorder (Eye disorders) | 0 | 0 | 0 | 1 (1)
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is an employee of the CRO who conducted the study and is restricted by CDA.

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT04932655/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04932655/SAP_001.pdf